CLINICAL TRIAL: NCT02226484
Title: Can Quercetin Increase Claudin-4 and Improve Esophageal Barrier Function in GERD?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nicholas Shaheen, MD, Professor of Medicine and Epidemiology Chief, Division of Gastroenterology & Hepatology, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-0557; 1R21DK097529-01A1 (NIH)
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Acid Reflux; Reflux
Keywords: Gastroesophageal reflux disease; GERD; Acid reflux; Reflux; Quercetin
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quercetin (Experimental): Two 250 mg capsules of oral quercetin (Q) twice-a-day (BID) one hour before meals with a glass of water for 6 weeks.
  Interventions: Drug: Quercetin

INTERVENTIONS:
Drug: Quercetin — Two 250 mg capsules of quercetin twice-a-day one hour before meals with a glass of water.

SUMMARY:
Purpose:

1. Determine if oral quercetin increases the expression of claudin-4 in the lining of the esophagus of patients with a diagnosis of gastroesophageal reflux disease (GERD); and
2. Determine whether the increase in claudin-4 by oral quercetin is accompanied by improvement in the barrier function and acid resistance of the lining of the esophagus of patients with a diagnosis of gastroesophageal reflux disease (GERD)

If interested, participants will be consented and provided a questionnaire to complete as part of the study. Participants will undergo endoscopy for routine care and will have up to 8 esophageal biopsies (small tissue samples) taken for the research study. After endoscopy, participants will be contacted to begin a 6 week treatment period with study drug (Quercetin, taken twice daily).

At the end of the 6 week period, participants will be scheduled to have blood drawn and to have a follow-up endoscopy with biopsies performed for the research study.

DETAILED DESCRIPTION:
Patients must be symptomatic (heartburn) and agree to allow endoscopic biopsies from the lower 5 cm of esophagus for research purposes. If the endoscopy demonstrates non-erosive reflux disease, biopsies of Esophageal Squamous Epithelium (ESE) are obtained and placed in mRNA-Later to assess claudin-4 mRNA by qRT-PCR and protein expression by Western blot (53, 64) while other biopsies of ESE are obtained and handled as in SpAim#2 to assess barrier function of ESE. After consent, subjects complete a questionnaire assessing demographics, disease-specific parameters such as duration of symptoms and past treatment, and the gastroesophageal reflux disease (GERD) Symptom Assessment Scale (GSAS), a validated measure of GERD severity. Following this, patients in open label fashion are given orally 500 mg Quercetin (Q) twice daily (bid) [Pure, House of Nutrition, Yonkers, NY] for 6-weeks. Symptoms are monitored 1 week before and for the 6 week treatment period. At 6 weeks, a blood sample is obtained for determination of Q and its metabolites by HPLC and endoscopy and biopsies of ESE are repeated and processed as initially done for claudin-4 levels in ESE.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to read, comprehend, and complete the consent form.
* Aged 18 to 80
* Diagnosed with gastroesophageal reflux disease (GERD) by a physician, defined as:

  a. History of heartburn at > 3 times/week for > 4 months AND either: i. Abnormal 24hr-pH monitoring (acid contact time > 4.5% OR ii. Past responsiveness to proton pump inhibitor (PPI) therapy
* Willing to undergo esophageal biopsy, endoscopy, and take study medication.
* Willingness to discontinue or remain off PPIs for the duration of the study (rescue medication use during the study such as antacids and H2 blockers as needed for symptoms is permitted)

Exclusion Criteria:

* Patients with a medical condition that makes him/her a poor risk for upper endoscopy, conscious sedation, esophageal biopsy or ability to comply with study directives
* Current use of blood thinners such as coumadin, warfarin, heparin and/or low molecular weight heparin, and rivaroxaban (requires discontinuation of medication 5 days prior to and 6 days after EGD)
* Patients with known bleeding disorders
* Patients who are status post partial or complete esophageal resection
* Patients with a history of esophageal or gastric surgery, includes fundoplication, gastric bypass, etc.
* Patients with a history of esophageal varices, esophageal cancer, achalasia, Barrett's esophagus, or eosinophilic esophagitis,
* Current diagnosis of invasive esophageal cancer
* Current use of calcium channel blockers, estradiol, immune suppressive drugs, aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), antibiotics, and/or taxol/paclitaxel
* Pregnant women
* Patients with a history of being intolerant of Quercetin
* Patients with continued moderate or severe heartburn despite use of twice daily PPIs (i.e. refractory to twice daily dosing of PPIs)
* Patients with current active erosive esophagitis (assessed during baseline EGD).
* Patients with a history of erosive esophagitis requiring PPI to treat. However, if patients have a history of erosive esophagitis and have discontinued PPI therapy at least 3 months prior to the baseline EGD, and there is no erosive disease seen during the baseline EGD, then these patients are eligible.
* Patients with significant erosive gastropathy on baseline EGD requiring PPI to treat clinically.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Expression of claudin-4 in esophageal squamous epithelium (ESE) of gastroesophageal reflux disease (GERD) in vivo | 6 weeks
  To assess the change in claudin-4 levels in a given subject before and after administration of Quercetin (Q), our null hypothesis is that there will be no difference in claudin-4 levels (i.e. mean Δ of claudin-4 titer from t0 to t1 is 0) and the alternative hypothesis is that claudin-4 levels following the administration of Q will be significantly different than before administration. To test this hypothesis, we will perform paired Student's t-tests. If data violate normality, Wilcoxon signed-rank test will be used as a nonparametric alternative to the Student's t. Additionally, exploratory analysis will be performed to assess the impact of treatment on reflux scores, as demonstrated by changes in the GERD Symptom Assessment Scale (GSAS) before and after therapy.

SECONDARY OUTCOMES:
Barrier function and acid resistance of esophageal squamous epithelium (ESE) as measured by epithelial resistance, RT, and fluorescein flux. | 6 weeks
  To determine whether the increase in claudin-4 by oral Quercetin (Q) is accompanied by improvement in the barrier function and acid resistance of esophageal squamous epithelium (ESE) in gastroesophageal reflux disease (GERD), we will assess the correlation in claudin-4 expression with our measures of epithelial resistance, RT, and fluorescein flux. Both the predictor variable (claudin-4 expression) and the response variables (RT and fluorescein flux) are continuous variables. Because the correlation between claudin-4 and the response variables is unknown and may not have a linear contour, Spearman's rank correlation coefficient will be used instead of Pearson's correlation, to improve sensitivity to non-linear relationships. Alpha will be set at 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data